CLINICAL TRIAL: NCT05554822
Title: Head-to-head Comparison of Single Versus Dual Antiplatelet Treatment Strategy After Percutaneous Left Atrial Appendage Closure: a Multicenter, Randomized Study - ARMYDA-AMULET
Brief Title: Head-to-head Comparison of Single Versus Dual Antiplatelet Treatment Strategy After Percutaneous Left Atrial Appendage Closure: a Multicenter, Randomized Study
Acronym: ARMYDA-AMULET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Giuseppe Patti, Scientific Director (Co-Chair), MD, Director, Chair of Cardiology, University of Eastern Piedmont, Novara; Director, Department of Thoracic and Cardiovascular Diseases, Maggiore della Carità Hospital, Novara, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-000730-34
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Left Atrial Appendage Occlusion; Antiplatelet Therapy
Keywords: left atrial appendage; left atrial appendage occlusion; atrial fibrillation; thromboembolic risk
MeSH Terms: conditions — Atrial Fibrillation | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single antiplatelet therapy (SAPT) (Experimental): Single antiplatelet therapy composed of aspirin 100 mg OD, organized as follows:
  Aspirin-naïve: aspirin 325 mg will be given 12-24 hours before the procedure and continued after the intervention at the dose of 100 mg OD up to 6-month follow-up.
  Aspirin-treated: periprocedural aspirin 100 mg OD will be given and continued up to 6-month followup.
  Interventions: Drug: Aspirin 100mg
- Double antiplatelet therapy (DAPT) (Active Comparator): Double antiplatelet therapy composed of aspirin 100 mg OD plus Clopidogrel 75 mg OD, organized as follows:
  Aspirin-naïve: aspirin 325 mg will be given 12-24 hours before the procedure and continued after the intervention at the dose of 100 mg OD up to 6-month follow-up. Clopidogrel will be given with a 300 mg loading dose of clopidogrel approximately 12 hours before the procedure and then clopidogrel 75 mg OD will be given from the day of intervention up to 3 months. At 3 months clopidogrel will be stopped.
  Aspirin-treated: periprocedural aspirin 100 mg OD will be given and continued up to 6-month followup. Clopidogrel will be given with a 300 mg loading dose of clopidogrel approximately 12 hours before the procedure and then clopidogrel 75 mg OD will be given from the day of intervention up to 3 months. At 3 months clopidogrel will be stopped.
  Interventions: Drug: Aspirin 100 mg OD plus clopidogrel 75 mg OD

INTERVENTIONS:
Drug: Aspirin 100mg — Single antiplatelet therapy with aspirin 100 mg OD for 6 months after the procedure
  Arms: Single antiplatelet therapy (SAPT)
Drug: Aspirin 100 mg OD plus clopidogrel 75 mg OD — Double antiplatelet therapy with Aspirin 100 mg OD plus clopidogrel 75 mg OD for 3 months, followed by 3 months of single antiplatelet therapy with aspirin 100 mg OD.
  Arms: Double antiplatelet therapy (DAPT)

SUMMARY:
The study will perform a randomized, head-to-head comparison between SAPT (aspirin) and DAPT (aspirin plus clopidogrel) after percutaneous LAA closure with implantation of the Amulet device (AbbottTM, Abbott Park, Illinois, US) in patients with AF. Primary outcome measure will be a net composite endpoint at 6 months including all-cause death, DRT, clinically relevant bleeding complications and ischemic events. The SAPT arm will receive aspirin alone up to 6 months, while the DAPT arm will receive DAPT for 3 months and then aspirin alone. Thus, between 3- and 6-month follow-up both groups will be given aspirin alone.

DETAILED DESCRIPTION:
State of the art There is no clear evidence on optimal antiplatelet therapy after percutaneous left atrial appendage (LAA) closure in patients with atrial fibrillation (AF). There is a consensus supporting dual antiplatelet therapy (DAPT) with aspirin plus clopidogrel (without oral anticoagulation) after non-WATCHMAN device implantation. However, the use of DAPT after LAA closure was initially derived from other interventional settings (e.g. the antithrombotic approach used after coronary stenting) and available data essentially derive from observational (and often retrospective), non-randomized, studies. Due to the lack of robust and consolidated evidence, the type and duration of antiplatelet therapy after LAA closure are variable and often guided by the individual convincement of the treating physicians. Patients undergoing LAA closure are generally older and have multiple co-morbidities; thus, in these patients the risk of bleeding events is a major concern and antithrombotic therapy may strongly contribute to such risk. Single-center, observational data have suggested that a strategy with single antiplatelet therapy (SAPT, essentially aspirin, without P2Y12 inhibitor) is associated with similar risk of ischemic cerebral events and device-related thrombosis (DRT) and with a significant reduction of bleeding complications after the intervention with 68% reduction in risk of major bleeding (from 7.0% to 2.3%). However, a recent, retrospective evidence raised concerns regarding the effectiveness of SAPT in preventing DRT in this setting of patients. To date, no randomized study has evaluated whether an approach with SAPT, compared to DAPT, is associated with adequate protection from DRT/ischemic events and with decreased bleeding risk. We will address such issue in a randomized, prospective, multicenter study.

Aim of the study The study will perform a randomized, head-to-head comparison between SAPT (aspirin) and DAPT (aspirin plus clopidogrel) after percutaneous LAA closure with implantation of the Amulet device (AbbottTM, Abbott Park, Illinois, US) in patients with AF. Primary outcome measure will be a net composite endpoint at 6 months including all-cause death, DRT, clinically relevant bleeding complications and ischemic events. The SAPT arm will receive aspirin alone up to 6 months, while the DAPT arm will receive DAPT for 3 months and then aspirin alone. Thus, between 3- and 6-month follow-up both groups will be given aspirin alone. We consider that a 6-month follow-up would be more than enough to detect any possible difference between the two groups.

Primary objective:

To demonstrate that SAPT is not inferior to the current standard antiplatelet therapy (DAPT) after LAA closure regarding the cumulative incidence of the net composite endpoint, including death, thrombotic complications and bleeding events, at 6 months.

Secondary objectives:

Compared to DAPT, SAPT use is associated with a similar incidence of ischemic events and a significantly lower incidence of bleeding complications at 6 months.

Study design The study will be phase IV, prospective, multicenter, with 1:1 randomization, open-label, with parallel groups. Consecutive patients with AF undergoing percutaneous LAA closure with the Amulet device will be enrolled. Patients will be included regardless of the type of AF and of clinical indication for LAA closure. Approximately 15 centers with a consolidated experience in the procedure of percutaneous LAA closure will be included. Enrollment will be competitive; each center will include a maximum number of patients corresponding to the 20% of the global population. After the protocol approval, the high-volume centers (e.g. top implanting centers in Italy) will be asked to participate the study, in addition to the Coordinating Center.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥18 years signing a specific informed consent
* Patients with a planned percutaneous LAA closure;
* Patients with documented non-valvular AF, irrespective of the type (paroxysmal, permanent, persistent), and CHA2DS2-VASc score ≥2
* Patients suitable for treatment with aspirin and clopidogrel according to the Summaries of product characteristics (SmPCs);
* Patients considered unsuitable for long-term oral anticoagulant therapy due to a high bleeding risk. Patients will be judged unsuitable for anticoagulation because of bleeding-prone comorbidities, history of previous bleeding (with or without anticoagulant treatment) or an expected low adherence to therapy.
* Patient's availability to undergo the follow-up visits scheduled for the study
* Negative pregnancy testing (if applicable), performed at the time of enrollment.

Exclusion Criteria:

* CHADS-VAsc score 0-1
* Requirement for on-going therapy with clopidogrel at the time of screening evaluation (e.g. current therapy with clopidogrel at the time of the screening evaluation will be an exclusion criterion)
* Known hypersensitivity to the study drugs (aspirin or clopidogrel)
* Patients deemed to be unsuitable for at least 6 months antiplatelet therapy (SAPT or DAPT) because of a recent (<1 month) major bleeding event
* Planned oral anticoagulant therapy after the procedure
* Moderate to severe mitral stenosis
* Mechanical heart prosthetic valve
* Active endocarditis
* Active bleeding
* Myocardial infarction or percutaneous coronary intervention <6 months
* Major surgery within one month
* Intracranial neoplasm, aneurysm or arterio-venous malformation
* Platelet count <50,000/μL
* Recent stroke (<1 month)
* Fibrinolytic therapy within 10 days
* Baseline hemoglobin <9 g/dL
* Pregnant woman
* Breast-feeding
* Women unavailable to use contraception during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint:all-cause death, DRT (at 3- or 6-month TEE), ischemic stroke, systemic embolic events (SEE) or BARC classification bleeding ≥3. | 6 months
  Primary endpoint will be the 6-month incidence in the two arms (SAPT versus DAPT) of the net composite endpoint including all-cause death, DRT (at 3- or 6-month TEE), ischemic stroke, systemic embolic events (SEE) or BARC classification bleeding ≥3. An independent board for clinical event adjudication and data safety monitoring will be created.

SECONDARY OUTCOMES:
Secondary endpoint: Device-related thrombosis | At 3 months and at 6 months
  Device-related thrombosis evaluated with transesophageal echocardiogram
Secondary endpoint: Any-cause death | 6 months
  Any-cause death
Secondary endpoint: ischemic stroke or systemic embolic events | At 3 months and at 6 months
  Incidence of ischemic stroke or systemic embolic events (SEE)
Secondary endpoint: Any bleeding | At 3 months and at 6 months
  Incidence of any bleeding
Secondary endpoint: BARC ≥3 bleeding | At 3 months and at 6 months
  Incidence of BARC classification bleeding ≥3

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Patti, MD, Study Director — University of Eastern Piedmont, Novara - Maggiore della Carità Hospital, Novara; Sergio Berti, MD, Principal Investigator — Fondazione Toscana G. Monasterio, Ospedale del Cuore "G. Pasquinucci"
Locations (19):
- Italy (19):
  - Azienda Ospedaliera Universitaria Policlinico Vittorio Emanuele Presidio Ospedaliero G. Rodolico, Catania
  - Presidi Ospedalieri Riuniti ASL 6 Ciriè - Presidio Ospedaliero Riunito Sede di Ciriè, Cirié
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Centro Cardiologico Fondazione Monzino, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera dei Colli Monaldi, Napoli
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Ospedale Maggiore della Carità, Novara
  - Clinica San Carlo, Paderno Dugnano
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Policlinico San Matteo, Pavia
  - Ospedale del Cuore G. Pasquinucci, Pisa
  - Ospedale di Rivoli, Rivoli
  - Ospedale S. Eugenio - ASL Roma 2, Roma
  - Azienda Ospedaliera Universitaria Sassari, Sassari
  - Ospedale Mauriziano Umberto I, Torino
  - Villa Maria Pia Hospital, Torino
  - Ospedale San Giovanni Bosco, Torino
  - Ospedale Sant'Andrea, Vercelli